CLINICAL TRIAL: NCT01845103
Title: Post-Approval Study of the PEARL 8.0 Handpiece for Transmyocardial Revascularization (TMR) With the Cardiogenesis Holmium:YAG Laser System
Brief Title: The PEARL 8.0 Post-Approval Study
Status: Terminated | Type: Observational
Why Stopped: Due to the product being discontinued
Sponsor: Cardiogenesis Corporation, a wholly-owned subsidiary of CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PLT1101.003-M
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Class IV Angina
Keywords: ANGINA; Thoracoscopic
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective single arm study of the Cardiogenesis PEARL 8.0 Handpiece Delivery System. The purpose of this study is to demonstrate that the 30 day mortality rate among patients who are treated with this device is less than the historical rate plus a non-inferiority margin.

DETAILED DESCRIPTION:
This is a prospective single arm study of the Cardiogenesis PEARL 8.0 Handpiece Delivery System. The PEARL 8.0 Handpiece allows the TMR laser energy to be directed at the heart through a small port up to 8 mm in size. The purpose of this study is to demonstrate that the 30 day mortality rate among patients who receive this device is less than the historical rate plus a non-inferiority margin. In a recent study of 34 patients treated with the PEARL 8.0 device, 3 (8.8%) experienced 30 day mortality. Among 132 patients in the original PMA trial treated with the SoloGrip III Handpiece, a similar device delivering identical energy, the 30 day mortality rate was 5.3% (7/132). In the Post-Approval Study of the SoloGrip III Handpiece, 2/72 prospectively enrolled patients died within the first 30 days. Therefore, the weighted average of the Pre-market and post-market studies has been calculated (4.4%) and will serve as the historical rate.

This trial will be monitored for success and futility according to a Bayesian adaptive design. Based on prior history, we assume patients will be accrued at the rate of approximately 1 patient per month and therefore, 30 day mortality will be known for all currently enrolled patients at the time each new patient is enrolled.

The success stopping boundaries for this study are 0/10 and 1/22. Thus, if no deaths are observed among the first 10 patients, the study will stop for success. If 1 death is observed among the first 10 patients, the study will continue to enroll. If among the first 22 patients, only 1 death is observed (there are no additional deaths), the study will stop for success. At any time, if 2 or more deaths are observed, the study will stop for futility.

A secondary objective is to assess the effect of channel number on the 30 day mortality rate to justify the labeling claims that the risk for early post-operative (30 day) mortality is associated with an increased number of channels, and not the function of the operation or device.

ELIGIBILITY:
Inclusion Criteria:

* Class IV angina (according to Canadian Cardiovascular Society Angina Scale)
* Ejection Fraction > 30%
* Patients with regions of myocardium in the distal two-thirds of the left ventricle with reversible ischemia and who are not eligible for direct coronary revascularization (e.g., CABG or PTCA).
* Patients amenable to thoracoscopic TMR.

Exclusion Criteria:

* Age less than18-years
* Pregnant or nursing mothers
* Unable to undergo a surgical procedure or general anesthesia
* Hepatic disease, renal failure, cancer or major infection
* Severely unstable angina (un-weanable from intravenous anti-anginals for 48- hours)
* Patients with mechanical/prosthetic heart valves
* Myocardial ischemia limited to the right ventricular wall
* Q-Wave myocardial infarction within three (3) weeks prior to the procedure
* Non Q-Wave myocardial infarction within two (2) weeks prior to the procedure
* Requires anticoagulation medications or has other hemorrhagic propensity
* Severe arrhythmia within one week prior to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of two and a maximum of five study sites will be selected for participation. The sites (surgeons) will be selected first from those that participated in the PEARL Study TMR 05-001. If additional sites are required, selection will be made for the sites (surgeons) to be familiar with TMR and thoracoscopic surgery. Sites will be asked to offer all patients eligible for stand-alone thoracoscopic TMR, who meet the inclusion/exclusion criteria, the opportunity to participate in the current study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Capps, MS, Study Director — CryoLife, Inc.
Locations (1):
- Sutter Institute for Medical Research, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PEARL 8.0: Received TMR with PEARL 8.0
Period: Overall Study
Arm/Group | PEARL 8.0
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PEARL 8.0
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Time Frame: 30 day
Measure: Number; unit: percentage of participants
Arm/Group | PEARL 8.0
Number analyzed (Participants) | 1
percentage of participants | 0

2. Secondary Outcome: Major Adverse Coronary and Cerebrovascular Events (MACCE)
Description: MACCE includes:
  Cardiac related death, CVA, Myocardial Infarction, Serious arrhythmia, CHF
Time Frame: 30 day
Measure: Number; unit: percentage of participants
Arm/Group | PEARL 8.0
Number analyzed (Participants) | 1
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | PEARL 8.0
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEARL 8.0 (N=1)
Serious Adverse Event required hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) — It was noted that this serious adverse event was not cardiac, procedural or device related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site and Investigator agree not to publish or present results prior to Sponsor's final report, but in no event shall Site or Investigator be restricted after the expiration of 12m from Project completion. Publication or disclosure made by Site or Investigator shall not contain Sponsor Confidential Information (CI) and text shall be submitted for Sponsor CI review and comment 30d prior to submission or disclosure and can be deferred, not exceeding 90d for the Sponsor to protect its rights in CI.